CLINICAL TRIAL: NCT00714870
Title: Pediatric Quality of Life Among Population With BMI Greater Than or Equal to 85%: Impact of a Behavioral Intervention Program
Brief Title: Pediatric Quality of Life Among Population With Body Mass Index (BMI) Greater Than or Equal to 85%
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steward St. Elizabeth's Medical Center of Boston, Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00446
Record Dates: First submitted 2008-07-09; First posted 2008-07-14 (Estimated); Results first posted 2013-05-31 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Pediatric Obesity
Keywords: BMI; Quality of life
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): intervention: this group will attend the nutrition and exercise program control group: this group will not attend the nutrition and exercise program
  Interventions: Behavioral: Behavioral nutrition and exercise program

INTERVENTIONS:
Behavioral: Behavioral nutrition and exercise program — The intervention consists of a behavioral nutrition and exercise program. Meetings occur monthly on a Saturday afternoon and last 4 hours. During this time we cover: 1)registration: monitoring of sedentary activities and liquid choices, motivational interviewing, exercise testing;2)exercise: includes strength training; 3) educational lectures; 4) didactic games and projects.

SUMMARY:
We are currently experiencing an epidemic of obesity in the Pediatric Population. This epidemic affects many areas including quality of life.

We have been conducting a nutrition and exercise program since 2003. We have noticed that many of the participants seem to have a better quality of life after finishing the one year program compared to when they started. We would like to objectively quantify this improvement using a validated questionnaire at the beginning and at the end of the study. Questionnaires will be given to participants and to their caretakers at the same time. There will be two groups in the study: one intervention (minimum attendance of 4 sessions) and one control group.

DETAILED DESCRIPTION:
We are currently experiencing an obesity epidemic in the Pediatric population. The latest National Health and Nutrition Examination Survey (NHANES) data indicates that 16.5% has a BMI greater than or equal to 85% < 95% and 17.1% has a BMI greater than or equal to 95%. The quality of life of children who are obese has been shown to be lower than that of children with cancer. Health related quality of life measurements have emerged as an important health outcome in clinical trials, clinical practice improvement strategies, and healthcare services research and evaluation. We have conducted a behavioral nutrition and exercise program since 2003. The name of the program is Teens, Empowerment, Exercise, Education, Nutrition (TEEEN) Program. We meet once a month on a Saturday afternoon for four hours. During this time we cover: registration (monitoring of sedentary activities and liquid choices; motivational interview, exercise testing); exercise; educational interactive lectures; didactic games and projects. We have noticed that participants seem to have a better quality of life after participating in the program compared to baseline. We would like to objectively quantify this subjective finding. We will be using the Pediatric Quality of Life Inventory Version 4.0 (PedsQL(TM)4.0) questionnaire which has been validated in the pediatric population. We will have an intervention and a control group. Both participants and their caretakers will be given a questionnaire at the beginning and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Ages 10-20
* BMI greater or equal to 85%

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2008-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Gonzalez, MD, Principal Investigator — Steward St. Elizabeth's Medical Center
Locations (1):
- Steward St. Elizabeth's Medical Center, Brighton, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with BMI % greater than or equal to 85% ages 9-20 were recruited from providers' offices between 2008-2012
Pre-assignment Details: Participants with endocrinologic conditions associated with weight gain were excluded from enrollment
Groups:
- Intervention: Nutrition and Exercise Program: intervention: this group will attend the nutrition and exercise program
  Behavioral nutrition and exercise program : The intervention consists of a behavioral nutrition and exercise program. Meetings occur monthly on a Saturday afternoon and last 4 hours. During this time we cover: 1)registration: monitoring of sedentary activities and liquid choices, motivational interviewing, exercise testing;2)exercise: includes strength training; 3) educational lectures; 4) didactic games and projects.
- Control Group: Standard of Care at Pediatrician's Office: control group: this group will not attend the nutrition and exercise program
Period: Overall Study
Arm/Group | Intervention: Nutrition and Exercise Program | Control Group: Standard of Care at Pediatrician's Office
Started | 49 | 27
Completed | 22 | 22
Not Completed | 27 | 5
Not completed — Lost to Follow-up | 22 | 5
Not completed — patient unable to come b/c back pain | 1 | 0
Not completed — did not attend minimum of 4 sessions | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Nutrition and Exercise Program: intervention: this group will attend the nutrition and exercise program control group: this group will not attend the nutrition and exercise program
  Behavioral nutrition and exercise program : The intervention consists of a behavioral nutrition and exercise program. Meetings occur monthly on a Saturday afternoon and last 4 hours. During this time we cover: 1)registration: monitoring of sedentary activities and liquid choices, motivational interviewing, exercise testing;2)exercise: includes strength training; 3) educational lectures; 4) didactic games and projects.
- Control Group: control group: this group will not attend the nutrition and exercise program
- Total: Total of all reporting groups
Arm/Group | Intervention: Nutrition and Exercise Program | Control Group | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21 | 22 | 43
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 11.6 (2.1) | 12 (2.3) | 11.8 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 20
  Male | 14 | 10 | 24
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Change in Child Self-report Health Related Quality of Life Scores After Intervention: Total, Physical and Psychosocial (Presented in This Order)
Description: Using a validated quality of life questionnaire we analyzed change in child self-report scores comparing baseline questionnaire scores to end of study questionnaire scores for these categories: total (includes physical and psychosocial), physical, and psychosocial(includes emotional, social, and school).
  Scale information: The range is 0-100 in terms of points they could get for each category. They had the options of 0-4, 0 being the best. 0 would then be transformed to a score of 100, 1 to 75, 2 to 50, 3 to 25 and 4 to 0.
  Results are clinically significant if the difference in scores are higher than the Minimal Clinical Important Difference (MCID). MCID are as follows: Total Score: 4.36, Physical Health: 6.66, Psychosocial Health: 5.30.
Time Frame: one year comparing change in questionnaire scores at baseline to results from questionnaire completed a year later
Population: To detect an effect with greater than or equal to 80% power at a 0.05 two sided significant level, we concluded we needed 22 participants completing each group, intervention and control
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control: Control group received the standard of care at pediatrician's office
Arm/Group | Intervention: Nutrition and Exercise Program | Control
Number analyzed (Participants) | 22 | 22
units on a scale
  Mean change in scores: Total | 7.8 (16.8) | -0.9 (15.6)
  Mean change in scores: Physical | 9.1 (22.5) | -0.3 (14.2)
  Mean change in scores: Psychosocial | 7.2 (17.7) | -1.2 (17.6)

ADVERSE EVENTS:
Time Frame: Adverse events were not collected
Arm/Group | Intervention: Nutrition and Exercise Program | Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes